CLINICAL TRIAL: NCT06658444
Title: Effect of Onion Extract Nanoparticle Gel Phonophoresis on Postsurgical Scar of Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, heba Haridy, lecturer of basic science department, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000114
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Scar; Previous Cesarean Section
MeSH Terms: conditions — Cicatrix | interventions — Phonophoresis

STUDY DESIGN:
Intervention Model Description: Ultrasound-based therapy has proven to be a viable option for treating abnormal scarring. It has been shown to reduce the growth of keloids or postoperative scars. Phonophoresis's advantages include noninvasiveness, good compliance, low cost, and minimal gastrointestinal side effects. Onion extracts were originally used for treating full and partial-thickness burns; however, more recently these have been trialed for treating hypertrophic and keloid scarring, and healing wounds. onion extract plays the main role in reducing scar through the inhibition of fibroblast proliferation and collagen production.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phonophoresis group (Experimental): Twenty women will receive onion extract phonophoresis (3 sessions/week) for 12 weeks in addition to deep friction massage.
  Interventions: Other: Phonophoresis
- control group (Sham Comparator): Twenty women will receive sham ultrasound (3 sessions/week) for 12 weeks in addition to deep friction massage.
  Interventions: Other: sham ultrasound

INTERVENTIONS:
Other: Phonophoresis — Pulsed ultrasound will be used at a frequency of 1 MHz with an intensity of 0.5 W/ cm2 for 5 minutes.
  Arms: phonophoresis group
Other: sham ultrasound — sham ultrasound
  Arms: control group

SUMMARY:
Cesarean section is one of the most common abdominal operations performed on women. The cesarean section rate is rising rapidly and continuously in many parts of the world. The cesarean-section surgery leaves a scar that requires special care. A horizontal skin incision approximately 10-15 cm long is usually performed during the procedure. Apart from the skin, the following: subcutaneous tissue, fascia, peritoneum, and uterine muscle are cut leaving traces in the form of scars and accompanying ailments, on the one hand, such as pain, tenderness, and hypersensitivity to stimuli, and on the other, limitations, such as contractures or impairment of tissue mobility

DETAILED DESCRIPTION:
All this may directly influence the patient's quality of life. There is also a significant negative impact on the psychological and social aspects of life, caused by the appearance of an unesthetic scar. Improper wound healing affects the area Therefore, it can affect the aesthetic appearance of the abdomen and cause, among others, posture asymmetry, gait disturbance, and pain in the lumbar spine. A growing number of patients are dissatisfied with the appearance of their scars. The efficacy of many existing prophylactic and therapeutic strategies has been proven through extensive use, also data on several approaches have been contradictory regarding the efficacy and side effects. Topical therapies have their advantages; specifically, increased adherence, the localized delivery of the product, and the reduced impact of first-pass metabolism. Onion extract contains a range of phenolic anti-oxidant and anti-inflammatory compounds and was originally used for treating full and partial-thickness burns; however, more recently these have been trialed for treating hypertrophic and keloid scarring, and healing wounds. onion extract plays the main role in reducing scars by inhibiting fibroblast proliferation and collagen production. onion extract is also believed to have anti-inflammatory and antimicrobial effects. Some studies on the preventive and treatment effectiveness of onion extract on hypertrophic scars demonstrated its capability to improve scar appearance Ultrasound-based therapy has shown to be a viable option for abnormal scarring. It has been shown to reduce the growth of keloids or postoperative scars and to facilitate the penetration of anti-scarring drugs into the dermis ). Advantages of phonophoresis include noninvasiveness, good compliance, low cost, and minimal gastrointestinal side effects

ELIGIBILITY:
Inclusion Criteria:

Their ages will be ≥18 years old. All women had given birth via elective abdominal transversal C-section for the first time.

All women suffering from Postsurgical Scar Of Cesarean-Section about 2-3 months post-surgery.

All women will provide an informed consent form agreeing to participate and publication of the study results

Exclusion Criteria:

Any pathological conditions or associated injuries affect the result of the study.

Skin disease. Cognitive and psychological impairment. Patients have implanted electronic devices, such as cardiac pacemakers, to prevent ultrasound interference.

Women with diabetes, cardiovascular problems, or a previous history of any disorder may alter sensation and delay the healing process which counteracts the study's goal.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Vancouver scar scale | 12 weeks
  Assesses four characteristics of vascularity, pigmentation, pliability, and height The larger the The larger the total score, the worse the scar . Normal skin (zero score)
Tonometer | 12 weeks
  Tonometer The measurement area is placed directly under the tissue tonometer. A blunt piston is pressed into the tissue by the weight, and the resulting output reading is shown. The measurements are proportional to the tissue's pliability. All measurement procedures will be explained to each woman in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Haridy, doctoral, Principal Investigator — Egypt
Locations (1):
- Heba, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No